CLINICAL TRIAL: NCT01798199
Title: VERVE* PROJECT: Study of the Acceptability of a Virtual Reality System on the Cognitive Stimulation of Patients With Alzheimer's Disease or Related Conditions. (*Vanquishing Apathy Through E-inclusion Using Realistic Virtual Environment)
Brief Title: Vanquishing Apathy Through E-inclusion Using Realistic Virtual Environment Project
Acronym: VERVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 12-PP-04
Record Dates: First submitted 2012-11-21; First posted 2013-02-25 (Estimated); Last update posted 2015-09-01 (Estimated); Status verified 2015-08

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer; virtual reality system; Alzheimer's disease related conditions
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Alzheimer disease (Experimental)
  Interventions: Other: The training by Verve System

INTERVENTIONS:
Other: The training by Verve System

SUMMARY:
Virtual environments and information communication technologies (ICT) offer large perspectives in the field of assistive care and rehabilitation.

As potentially endless, the scenarios and environment used using 3D can provide immersive social and interactive context for enjoyable and therapeutic exercises in the aging population. In addition it is also possible to use this type of serious game and scenario in very easy to use devices such as lap top or tablet.

Social exclusion has many causes, Apathy as one of the most common behavioural disturbances found in old adults populations alters significantly social and emotional interaction.

Even though, progress in VR has been made over the past year, the presence of such technology in daily living space is still at the embryonic stage.

The European e-Inclusion policy stresses the importance of ICT in improving the quality of life in potentially disadvantaged groups, including older people and persons.

The VERVE project is developing ICT tools to support the treatment of people who are at risk of social exclusion due to apathy associated with a disability.

As people aged and autonomy worsen fear for safety and comfortable means to maintain social and Health Related Quality of Life (HRQL) status are public health issues.

Moreover, even though older adults would like to perform some activities such as walking in the streets some are reluctant to go out of their homes as the external environment is perceived as potentially unsafe.

Apathy, the most common behavioural symptoms in aging population is characterized by symptoms of reduced initiation and responsiveness to environmental interactions. The syndrome of Apathy takes form of diminished goal-directed behaviour, characterised by emotional blunting, loss of initiative and loss of interest. Apathy along with the nosological characteristics of dementia induces impairment in autonomy level and therefore dependence as cognitive impairments worsened.

The importance of stimulation could be related to the concept of engagement defined as the act of being occupied or involved with an external stimulus. Engaging older person with or without Alzheimer's disease and related disorders in appropriate activities has been shown to yield beneficial HRQL effects such increasing positive emotion, improving cognition, functional autonomy and quality of life.

Accordingly, enriched environments with high definition virtual representation of cities and activities of interest have the potentials not only to encourage patients to get active in a safe and interactive environment but also to create access to enjoyable and stimulating settings for the more severe patients.

The VR setting from VERVE proposed personalised and populated environments available on two different, but interlinked hardware platforms: 1/: standard gaming set-up in the home, nursing home or day hospital therapy group; and 2/ mobile tracked internet devices (e.g.,IPad). The system will ensure maximum openness and dissemination by using 3D Web technologies.

ELIGIBILITY:
Inclusion Criteria to MILD COGNITIVE IMPAIRMENT:

* Male or Female aged ≥ 60 years.
* Subject presenting a diagnosis of MCI according to the criteria of the National Institute on Aging and Alzheimer Association group (Albert M.S., 2011) ; or Alzheimer disease at the prodromal stage (Dubois B., 2010 )
* Subject presenting a score of 0 at the " Tremor " and " Rigidity " items from the UPDRS III
* Patient not presenting a major depression episode according to the DSM IV-R;
* Be affiliate to the social security system (For French patients only);
* Case of patients under guardianship after agreement of the guardian (legal entity);
* Signed and dated a written informed consent obtained from the subject

Exclusion Criteria to MILD COGNITIVE IMPAIRMENT:

-

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2013-05; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
the participants and careers acceptability | 8 weeks
  The primary objective is to evaluate the participants and careers acceptability in short and long term use of the VERVE light portable system used for cognitive stimulation of patients with cognitive pathologies.

SECONDARY OUTCOMES:
To assess the impact of behavioral disturbances over the use of the VR using the NPI and the Apathy Inventory | at 3, 4 and 8 weeks
  To assess the impact of behavioral disturbances over the use of the VR using the NPI and the Apathy Inventory
To describe the parameters those facilitate engagement within the designs of VERVE VR setting using the engagement scale OME | at 1, 2, 3, a weeks
  To describe the parameters those facilitate engagement within the designs of VERVE VR setting using the engagement scale OME
To assess the potential acceptability and preventive effectiveness of such setting in home setting using visual analogic scale and EQ-D6 | at 3, 4, 8 weeks
  To assess the potential acceptability and preventive effectiveness of such setting in home setting using visual analogic scale and EQ-D6
To assess cognitive impact of the light VERVE setting. Using Stroop, TMT, VAT and functional task (IADL) | First day and 4 weeks
  To assess cognitive impact of the light VERVE setting. Using Stroop, TMT, VAT and functional task (IADL)

CONTACTS AND LOCATIONS:
Overall Officials: Philippe ROBERT, PU-PH, Study Director — Centre Hospitalier Universitaire de Nice; Renaud DAVID, PH, Study Chair — CHU NICE; Guillaume SACCO, PH, Study Chair — Centre Hospitalier Universitaire de Nice; Jean Michel TURPIN, PH, Study Chair — Centre Hospitalier Universitaire de Nice
Locations (3):
- France (3):
  - CHU de Nice, Nice
  - EHPAD Valrose, Nice
  - EHPAD Villa Hélios Saint Jean, Nice